CLINICAL TRIAL: NCT01279733
Title: Prenatal Cytogenetic Diagnosis by Array-Based Copy Number Analysis
Acronym: Microarray
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ronald J Wapner, MD, Professor of Obstetrics & Gynecology, Columbia University
Other Study IDs: AAAC8036; 1R01HD055651-01 (NIH)
Record Dates: First submitted 2010-07-19; First posted 2011-01-19 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Genetic Diseases
Keywords: microarray
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Microarray Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Additional 15 ml of amniotic fluid (minimum 10 ml) for amniocentesis
  * Blood sample (10 ml) from each parent will be obtained in case of a need to test for suspected familial copy number variants (CNVs) or discrepant results, and also to evaluate for maternal cell contamination (patient's blood sample).
  * 10 ml of amniotic fluid with suspended cells, (minimum 7 ml)
  * 5 mg of villi (minimum of 2mg)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Microarray Analysis
  Interventions: Genetic: Microarray analysis

INTERVENTIONS:
Genetic: Microarray analysis — Microarray performed on prenatal specimen:
  Fluorescence in-situ hybridization (FISH) or other standardized tests such as qPCR or MLPA will be performed on the fetal sample to confirm abnormal MA findings of known and unknown clinical significance which are discordant with CC findings, including anomalies normally detected by karyotyping.
  Microarray analysis of DNA from parental blood samples will be used to determine whether CNVs detected in a fetal sample are also present in a healthy parent, in which case no further evaluation will take place, moreover any finding in a fetus which is duplicated in a parental microarray is considered to be confirmed.

SUMMARY:
The main objective of the multi-centered collaborative study is to evaluate the accuracy, efficacy and clinical advantages of prenatal diagnosis using microarray analysis as compared with conventional karyotyping.

DETAILED DESCRIPTION:
Specifically, the aims are as follows:

1. Demonstrate the performance of microarray analysis as a clinical method for prenatal cytogenetic diagnosis with regard to:

   1. Accuracy in the detection of the common autosomal and sex chromosomal aneuploid (trisomies, 13,18,21, 45,X, 47,XXY, etc.)
   2. Ability of microarray to diagnose less common, but clinically significant, cytogenetic aneusomies (e.g. DiGeorge, Williams, Smith- Magenis, Prader-Willi syndrome, etc.) currently not detected by conventional karyotype.
   3. Evaluation of the utility of microarray in specific clinical scenarios such as ultrasound detection of congenital anomalies and fetal growth disorders.
2. Evaluate the appropriate construction of prenatal diagnostic microarray devices to allow maximal detection of clinically relevant information with minimal detection of unexpected and difficult to interpret findings which have no clinical significance but might provoke patient anxiety.
3. Evaluate the feasibility and cost-effectiveness of using microarrays as a primary prenatal diagnostic tool.
4. Evaluate approaches to integrate microarray into clinical prenatal cytogenetic diagnostic practice.
5. Develop a prenatal diagnostic tissue repository (TDR) to facilitate the further development of microarray technology. This will be used to investigate the molecular etiologies of specific fetal anomalies and to test newer technologies, such as higher resolution microarrays.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy having either chorionic villus sampling in the first trimester or an amniocentesis procedure at or after 16 weeks of gestation performed for prenatal cytogenetic diagnosis
2. Karyotyping to be performed at Genzyme Genetics Cytogenetics Laboratory
3. Trained study personnel available
4. Presenting at pre-specified sites using Genzyme Genetics for routine prenatal diagnostic services

Exclusion Criteria:

1. Unavailability of one or both biologic parents to provide blood sample (e.g. egg or sperm donor, non-paternity)
2. Patient refusal to allow follow-up through the neonatal period and up to age two if selected
3. Participation in the study in a previous pregnancy
4. Insufficient sample for microarray assay

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 4,400 prenatal diagnostic samples will be obtained from patients undergoing prenatal testing for standard indications. Patients will be recruited at participating prenatal diagnostic centers by designated study personnel; recruitment of patients will be initiated as a pilot study. These patients will not contribute to the final planned sample size of 4400 patients. Two sub-studies will then be initiated consisting of 250 (or more) patients enrolled with sufficient amniotic fluid sample and 250 (or more) patients with sufficient villus sample.
Sampling Method: Non-Probability Sample
Enrollment: 4450 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Detection rate of fetal cytogentic abnormalites between microarray copy number analysis and karyotype in prenatal samples | Up to 2.5 years after recruitment of 4400 patients.
  This is a blinded prospective comparison of microarray copy number analysis to metaphase karyotyping for the detection of common fetal cytogentic abnormalites

SECONDARY OUTCOMES:
The ability of microarray copy number analysis to identify clinically significant microdeletions and duplications not seen by standard karyotyping | Up to 2.5 years .
  This outcome will identify the frequency of clinically significant microdeletions and microduplications that are identified on microarray CNA that were not seen on the clinical karyotype. Only copy number variants over 1 Mb in the backbone and those in predesignated critical regions will be included
The rates of clinically significant copy number variants associated with specific prenatal conditions | Up to 2.5 years after recruitment of 4400 patients.
  THe frequency of clinically significant copy number variants in cases with fetal anomalies, advanced maternal age, positve serum screening, and fetal growth disorders will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wapner, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Wapner RJ, Martin CL, Levy B, Ballif BC, Eng CM, Zachary JM, Savage M, Platt LD, Saltzman D, Grobman WA, Klugman S, Scholl T, Simpson JL, McCall K, Aggarwal VS, Bunke B, Nahum O, Patel A, Lamb AN, Thom EA, Beaudet AL, Ledbetter DH, Shaffer LG, Jackson L. Chromosomal microarray versus karyotyping for prenatal diagnosis. N Engl J Med. 2012 Dec 6;367(23):2175-84. doi: 10.1056/NEJMoa1203382. PMID 23215555